CLINICAL TRIAL: NCT02449044
Title: International, Multicenter, Study of One-year, Open-label, Titrated Oral Tolvaptan Tablet Administration in Patients With Chronic Hyponatremia: Extension to Studies 156-02-235 and 156-03-238 to Assess One-year Safety
Brief Title: International, Multicenter, Study of One-year, Open-label, Titrated Oral Tolvaptan Tablet Administration in Patients With Chronic Hyponatremia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-03-244
Record Dates: First submitted 2015-05-14; First posted 2015-05-20 (Estimated); Results first posted 2016-01-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Hyponatremia
Keywords: Hyponatremia
MeSH Terms: conditions — Hyponatremia | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tolvaptan (Experimental): Enrolled subjects began treatment with 15 mg tolvaptan QD. A titration between target doses of 15 mg, 30 mg, or 60 mg of trial medication was based on the subject's change in serum sodium concentration and clinical tolerance of the trial medication.
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — Once Daily

SUMMARY:
This study will assess the safety of long-term tolvaptan use in patients previously enrolled in shorter-term Phase 3 studies and gather information on the natural history of hyponatremia in the context of tolvaptan therapy and underlying disease states.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years.
2. Ability to provide informed consent or assent.
3. Prior successful participation in a tolvaptan hyponatremia trial termination with evidence of continued need or desire for therapy.

Exclusion Criteria:

* A current medical condition where long-term treatment with an aquaretic agent may present an undue risk to the patient.
* Hyponatremia which is acute, reversible, artifactual or due to conditions not associated with vasopressin excess or likely to respond to aquaretic therapy.
* Hyponatremia due to reversible medical condition or therapy
* Conditions associated with an independent imminent risk of morbidity and mortality
* Conditions which confound the assessment of endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2004-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

REFERENCES:
- [Result] Berl T, Quittnat-Pelletier F, Verbalis JG, Schrier RW, Bichet DG, Ouyang J, Czerwiec FS; SALTWATER Investigators. Oral tolvaptan is safe and effective in chronic hyponatremia. J Am Soc Nephrol. 2010 Apr;21(4):705-12. doi: 10.1681/ASN.2009080857. Epub 2010 Feb 25. PMID 20185637

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 111 enrolled participants at 33 trial centers. This is an extension study of trials NCT00072683 and NCT00201994. Approximately 50% participants may have been on tolvaptan previously, there was a minimum 7-day period off treatment between trials.
Pre-assignment Details: Participants were blinded prior to treatment with tolvaptan with titration between target doses of 15mg, 30mg or 60mg of study drug was based on the participant's response in serum sodium concentration and clinical tolerance of study drug. Dose titration aim was to stabilize the participants with normal range of blood sodium.
Groups:
- Tolvaptan: Participants received 15 mg tolvaptan QD and were titrated from 15mg, 30mg, or 60mg of tolvaptan based on the participant's response in serum sodium concentration and clinical tolerance of study drug.
Period: Overall Study
Arm/Group | Tolvaptan
Started | 111
Completed | 47 (Participants who completed Weeks 58, 106 and 216 visit.)
Not Completed | 64
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 13
Not completed — Adverse Event | 30
Not completed — Met Withdrawal Criteria | 7
Not completed — Physician Decision | 9
Not completed — Sponsor Discontinued Trial | 3

BASELINE CHARACTERISTICS:
Arm/Group | Tolvaptan
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 55

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Events (AEs)
Description: A TEAE was an AE that began after the first injection or was continuous from Baseline and was defined as any new medical problem, or exacerbation of an existing problem, whether or not it was considered drug-related by the study physician. An AE was considered serious if it was fatal; life-threatening; persistently or significantly disabling or incapacitating; required in-subject hospitalization or prolonged hospitalization; a congenital anomaly/birth defect; or other medically significant event that, based upon appropriate medical judgment, may have jeopardized the participant and may have required medical or surgical intervention to prevent the outcomes mentioned above.
Time Frame: Baseline to Post-Week 214 follow-up visit
Population: The ITT dataset, which comprised of data from all enrolled participants who had observations at Baseline and at least one Post-Baseline visit, were analyzed.
Measure: Number; unit: participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 111
participants
  Participants with TEAEs | 105
  Participants with serious TEAEs | 76
  Participants with severe TEAEs | 73
  Participants discontinued IMP due to TEAE | 19
  Participants discontinued IMP due to TEAE/death | 28
  Deaths | 19

2. Primary Outcome: Participants With Laboratory Values Abnormalities Reported as TEAEs
Description: The laboratory values were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal values in serum chemistry, hematology, urinalyses and prolactin tests that were identified based on pre-defined criteria. Any value outside the normal range was flagged for the attention of the study physician who was to indicate whether the value was clinically significant for identifying laboratory values of potential clinical relevance. Participants noted with abnormal laboratory values are reported below.
Time Frame: Baseline to Post-Week 214 follow-up visit
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 111
participants
  Serum Chemistry-Blood creatinine increased | 4
  Serum Chemistry-Blood potassium increased | 4
  Serum Chemistry-Blood glucose increased | 3
  Serum Chemistry-Blood potassium decreased | 3
  SerumChemistry-Aspartate aminotransferaseincreased | 2
  Serum Chemistry-Blood cholesterol increased | 3
  Serum Chemistry-Blood sodium increased | 2
  Serum Chemistry-Hepatic enzyme increased | 2
  Serum Chemistry-Oxygen saturation decreased | 2
  Serum Chemistry-Hyperglycaemia | 5
  Serum Chemistry-Hyperkalaemia | 7
  Serum Chemistry-Hyperlipidaemia | 4
  Serum Chemistry-Hypernatraemia | 4
  Serum Chemistry-Hyperuricaemia | 3
  Serum Chemistry-Hypoglycaemia | 5
  Serum Chemistry-Hypokalaemia | 14
  Serum Chemistry-Hypomagnesaemia | 3
  Serum Chemistry-Hypoatraemia | 25
  Hematology-Anemia | 20
  Hematology-Thrombocytopenia | 2
  Hematology-International normalized ratioincreased | 4
  Hematology-White blood cell count increased | 2

3. Primary Outcome: Participants With Electrocardiogram (ECG) Related Abnormalities Reported as TEAEs
Description: The ECG was one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance included abnormal values in HR outliers, PR outliers, QRS outliers, QT, QTcB, QTcF that were identified based on pre-defined criteria. Some of the pre-defined criteria for identifying ECG measurements of potential clinical relevance included: For QTcB and QTcF: baseline mean of QTcB and QTcF interval was new onset >500 msec, 30 - 60 msec, >60 msec; For QT: new onset >500 msec; For QRS outliers: >=25% change from baseline when QRS >100 msec; PR outliers: >=25% change from baseline when PR>200 msec; HR outliers: 25% decrease from baseline and HR <50 bpm or 25% increase from baseline and HR >100 bpm. New onset (>500 msec) in QT, QTcB, or QTcF means a participant who attained a value >500 msec during treatment period but not at each baseline visit. The ECG-related abnormalities are reported as TEAEs are mentioned below.
Time Frame: Baseline to Post-Week 214 follow-up visit
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 111
participants
  Atrial fibrillation | 6
  Tachycardia | 4
  Atrial tachycardia | 3
  First degree atrioventricular block | 2
  Bradycardia | 2
  Sinus tachycardia | 2
  Ventricular tachycardia | 2
  Left bundle branch block | 1
  Tachyarrhythmia | 1
  Ventricular arrhythmia | 1
  Atrial flutter | 1
  ECG ST segment depression | 1
  Arrhythmia | 1

4. Primary Outcome: Participants With Vital Signs Abnormalities Reported as Treatment Emergent Adverse Events (TEAEs)
Description: The vital signs were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance included abnormal values in body temperature, heart rate, systolic and diastolic blood pressure, respiratory rate and weight that were identified based on pre-defined criteria. Criteria for identifying vital signs of potential clinical relevance included: Heart rate, supine: >= 120 beats per minute (bpm) + increase of ≥15 bpm from Baseline and <=50 bpm + decrease of >= 15 bpm; Diastolic Blood Pressure, Supine: >=105 mmHg + increase of >=15 mmHg and <=50 mmHg + decrease of >=15 mmHg; Systolic Blood Pressure, Supine: >=180 mmHg + increase of >=20 mmHg and <= 90 mmHg + decrease of >=20 mmHg; Temperature (degree C): Increase of >=1.1 to >=38.3C. The vital sign abnormalities were reported as TEAEs are mentioned below.
Time Frame: Baseline to Post-Week 214 follow-up visit
Population: The intent-to-treat (ITT) dataset, which comprised of data from all enrolled participants who had observations at Baseline and at least one Post-Baseline visit, were analyzed.
Measure: Number; unit: participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 111
participants
  Hypotension | 13
  Hypertension | 8
  Pyrexia | 6
  Increased body temperature | 3
  Palpitations | 2
  Increased central venous pressure | 2
  Increased venous pressure | 1
  Orthostatic hypotension | 1
  Hypertensive crisis | 1
  Decreased orthostatic blood pressure | 1
  Increased weight | 5
  Decreased weight | 1

5. Primary Outcome: Participants With Body Weight Abnormalities Reported as TEAEs
Description: The body weight evaluation was one of the primary parameters to measure the safety and tolerability of individual participants. Every effort was made to ensure that body weight measurements were performed in a reproducible and consistent manner. The pre-defined criteria was change of ≥7% in body weight for both male and female. Participants were to wear the same type of clothes at each measurement, preferably a gown and no shoes. All body weight measurements were to have been taken post-void.
Time Frame: Baseline to Post-Week 214 follow-up visit
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 111
participants
  Increased weight | 5
  Decreased weight | 1

6. Secondary Outcome: Mean Change From Baseline in Serum Sodium Measurements
Description: Sodium measurements obtained at designated intervals were compared to each participant's Baseline sodium level at the beginning of placebo-controlled therapy in their original trial and from Baseline on initiation of therapy in the open-label trial.
Time Frame: Baseline of parent trial to Week 214
Population: The ITT dataset, which comprised of data from all enrolled participants who had observations at Baseline and at least one Post-Baseline visit, were analyzed. In the last observation carried forward (LOCF) dataset, missing data were filled in using the participant's preceding non-missing value, except that Baseline value will not be carried forward.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Tolvaptan
Number analyzed (Participants) | 111
mEq/L
  Day 1 post-dose (N= 99) | 2.2 (3.3)
  Day 14 (N= 110) | 5.2 (5.5)
  Day 31 (N= 110) | 5.0 (4.8)
  Week 10 (N= 110) | 5.0 (5.1)
  Week 18 (N= 110) | 4.6 (5.4)
  Week 26 (N= 110) | 4.2 (5.7)
  Week 34 (N= 110) | 4.7 (5.9)
  Week 42 (N= 110) | 5.2 (5.6)
  Week 50 (N= 110) | 5.0 (5.9)
  Week 58 (N= 110) | 5.0 (5.9)
  Week 70 (N= 110) | 4.8 (5.8)
  Week 82 (N= 110) | 4.8 (5.7)
  Week 94 (N= 110) | 5.1 (5.8)
  Week 106 (N= 110) | 5.0 (6.0)
  Week 118 (N= 110) | 4.8 (5.9)
  Week 130 (N= 110) | 4.9 (6.0)
  Week 142 (N= 110) | 5.2 (5.9)
  Week 154 (N= 110) | 5.2 (5.9)
  Week 166 (N= 110) | 4.9 (5.8)
  Week 178 (N= 110) | 4.8 (5.9)
  Week 190 (N= 110) | 5.1 (6.1)
  Week 202 (N= 110) | 5.0 (5.9)
  Week 214 (N= 110) | 5.0 (5.9)
Statistical Analysis 1: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Day 1
Statistical Analysis 2: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Day 14
Statistical Analysis 3: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Day 31
Statistical Analysis 4: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 10
Statistical Analysis 5: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 18
Statistical Analysis 6: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 26
Statistical Analysis 7: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 34
Statistical Analysis 8: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 42
Statistical Analysis 9: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 50
Statistical Analysis 10: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 58
Statistical Analysis 11: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 70
Statistical Analysis 12: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 82
Statistical Analysis 13: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 94
Statistical Analysis 14: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 106
Statistical Analysis 15: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 118
Statistical Analysis 16: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 130
Statistical Analysis 17: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 142
Statistical Analysis 18: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 154
Statistical Analysis 19: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 166
Statistical Analysis 20: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 178
Statistical Analysis 21: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 190
Statistical Analysis 22: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 202
Statistical Analysis 23: Comparison: Tolvaptan; Test type: Superiority or Other; p < 0.0001, Student's t-test — This was the p-value for analysis at Week 214

7. Secondary Outcome: Change From Baseline in Percentage of Participants With Severe Hyponatremia
Description: Percentage of participants with varying degrees of hyponatremia ("severe" <130, "mild" 130-135, "normal" >135 mEq/L) at Baseline and each study visit.
Time Frame: Baseline to Week 214
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 111
percentage of participants
  Day 1 post-dose (N=99) | 20.2 (3.0)
  Day 31 (N=110) | 9.1 (5.1)
  Week 10 (N=110) | 11.8 (5.0)
  Week 18 (N=110) | 13.6 (4.0)
  Week 26 (N=110) | 16.4 (4.6)
  Week 34 (N=110) | 14.5 (5.6)
  Week 42 (N=110) | 12.7 (4.1)
  Week 50 (N=110) | 10.9 (4.5)
  Week 58 (N=110) | 13.6 (5.1)
  Week 70 (N=110) | 12.7 (4.6)
  Week 82 (N=110) | 10.9 (4.1)
  Week 94 (N=110) | 10.9 (4.8)
  Week 106 (N=110) | 12.7 (4.7)
  Week 118 (N=110) | 12.7 (4.4)
  Week 130 (N=110) | 11.8 (4.7)
  Week 142 (N=110) | 11.8 (4.5)
  Week 154 (N=110) | 11.8 (4.4)
  Week 166 (N=110) | 11.8 (4.5)
  Week 178 (N=110) | 11.8 (4.5)
  Week 190 (N=110) | 11.8 (4.7)
  Week 202 (N=110) | 11.8 (4.6)
  Week 214 (N=110) | 11.8 (4.6)

8. Secondary Outcome: Change From Baseline in Percentage of Participants With Mild Hyponatremia
Description: as for outcome 7
Time Frame: Baseline to Week 214
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 111
percentage of participants
  Day 1 post-dose (N=99) | 53.5
  Day 31 (N=110) | 33.6
  Week 10 (N=110) | 28.2
  Week 18 (N=110) | 33.6
  Week 26 (N=110) | 30.9
  Week 34 (N=110) | 26.4
  Week 42 (N=110) | 26.4
  Week 50 (N=110) | 31.8
  Week 58 (N=110) | 26.4
  Week 70 (N=110) | 30.9
  Week 82 (N=110) | 31.8
  Week 94 (N=110) | 28.2
  Week 106 (N=110) | 27.3
  Week 118 (N=110) | 28.2
  Week 130 (N=110) | 29.1
  Week 142 (N=110) | 25.5
  Week 154 (N=110) | 25.5
  Week 166 (N=110) | 30.9
  Week 178 (N=110) | 30.9
  Week 190 (N=110) | 30.9
  Week 202 (N=110) | 30.9
  Week 214 (N=110) | 30.9

9. Secondary Outcome: Change From Baseline in Percentage of Participants With Normal Sodium Levels
Description: as for outcome 7
Time Frame: Baseline to Week 214
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 111
percentage of participants
  Day 1 post-dose (N=99) | 26.3
  Day 31 (N=110) | 57.3
  Week 10 (N=110) | 60.0
  Week 18 (N=110) | 52.7
  Week 26 (N=110) | 52.7
  Week 34 (N=110) | 59.1
  Week 42 (N=110) | 60.9
  Week 50 (N=110) | 57.3
  Week 58 (N=110) | 60.0
  Week 70 (N=110) | 56.4
  Week 82 (N=110) | 57.3
  Week 94 (N=110) | 60.9
  Week 106 (N=110) | 60.0
  Week 118 (N=110) | 59.1
  Week 130 (N=110) | 59.1
  Week 142 (N=110) | 62.7
  Week 154 (N=110) | 62.7
  Week 166 (N=110) | 57.3
  Week 178 (N=110) | 57.3
  Week 190 (N=110) | 57.3
  Week 202 (N=110) | 58.2
  Week 214 (N=110) | 57.3

10. Secondary Outcome: Percentage of Participants Requiring Prescription of Fluid Restriction
Description: Percentage of participants requiring prescription of fluid restriction for the express purpose of treating hyponatremia during each period of the trial. Assessed descriptively at each visit.
Time Frame: Baseline to Post-Week 214 follow-up visit
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 111
percentage of participants
  Mild Hyponatremia (N=76) | 14.47
  Severe Hyponatremia (N=35) | 5.71

11. Secondary Outcome: Number of Participants Requiring Prescription of Hypertonic Saline
Description: Percentage of participants requiring prescription of hypertonic saline for the express purpose of treating hyponatremia during each period of the trial, assessed descriptively at each visit.
Time Frame: Baseline to Post-Week 214 follow-up visit
Population: The ITT dataset, which comprised of data from all enrolled participants who had observations at Baseline and at least one Post-Baseline visit, were analyzed. Percentage of participants requiring prescription of hypertonic saline was not analyzed due to a low number of participants who received the treatment.
Measure: Number; unit: participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 111
participants | 2

12. Secondary Outcome: Percentage of Participants Requiring Prescription of Other Medicines
Description: Percentage of participants requiring prescription of other medicines for the express purpose of treating hyponatremia during each period of the trial, assessed descriptively at each visit.
Time Frame: Baseline to Post-Week 214 follow-up visit
Population: The ITT dataset, which comprised of data from all enrolled participants who had observations at Baseline and at least one Post-Baseline visit, were analyzed. Percentage of participants requiring other medicines such as demeclocycline or urea was not analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 111
percentage of participants | 0

13. Secondary Outcome: Mean Change From Baseline in Body Weight by Visit for Those Participants Who Had Clinical Evidence of Hypervolemia at Baseline
Description: Body weight at each visit (assessed only for those with clinical evidence of hypervolemia at Baseline) and was summarized using descriptive statistics.
Time Frame: Baseline to Week 214
Population: The ITT dataset comprised of data from all enrolled participants who had observations at Baseline and at least one Post-Baseline visit were analyzed. The observed cases (OC) dataset consisted of only data points obtained from participants who were evaluated at the visit, without missing study drug consecutively for 14 days.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Tolvaptan
Number analyzed (Participants) | 111
kg
  Day 31 (N= 26) | -0.5 (4.6)
  Week 10 (N= 32) | -1.1 (3.7)
  Week 18 (N= 27) | 0.2 (3.0)
  Week 26 (N= 27) | 0.4 (5.4)
  Week 34 (N= 26) | 0.5 (4.0)
  Week 42 (N= 24) | 0.3 (4.6)
  Week 50 (N= 22) | 1.0 (4.7)
  Week 58 (N= 22) | 1.7 (4.5)
  Week 70 (N= 18) | 1.7 (5.2)
  Week 82 (N= 18) | 2.0 (7.0)
  Week 94 (N= 18) | 3.0 (8.0)
  Week 106 (N= 15) | 1.4 (8.0)
  Week 118 (N= 13) | 2.2 (8.1)
  Week 130 (N= 13) | 3.0 (9.0)
  Week 142 (N= 12) | 3.8 (8.7)
  Week 154 (N= 11) | 2.7 (7.9)
  Week 166 (N= 9) | 2.9 (9.4)
  Week 178 (N= 7) | 3.2 (8.6)
  Week 190 (N= 5) | -2.4 (4.5)
  Week 202 (N= 2) | -7.1 (0.4)
  Week 214 (N= 2) | -8.5 (1.6)
Statistical Analysis 1: Comparison: Tolvaptan; Statistical analysis at Day 31; Test type: Superiority or Other; p = 0.4922, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 2: Comparison: Tolvaptan; Statistical analysis at Week 10; Test type: Superiority or Other; p = 0.1054, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 3: Comparison: Tolvaptan; Statistical analysis at Week 18; Test type: Superiority or Other; p = 0.7656, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 4: Comparison: Tolvaptan; Statistical analysis at Week 26; Test type: Superiority or Other; p = 0.7084, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 5: Comparison: Tolvaptan; Statistical analysis at Week 34; Test type: Superiority or Other; p = 0.5138, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 6: Comparison: Tolvaptan; Statistical analysis at Week 42; Test type: Superiority or Other; p = 0.7175, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 7: Comparison: Tolvaptan; Statistical analysis at Week 50; Test type: Superiority or Other; p = 0.3540, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 8: Comparison: Tolvaptan; Statistical analysis at Week 58; Test type: Superiority or Other; p = 0.0852, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 9: Comparison: Tolvaptan; Statistical analysis at Week 70; Test type: Superiority or Other; p = 0.1923, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 10: Comparison: Tolvaptan; Statistical analysis at Week 82; Test type: Superiority or Other; p = 0.2335, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 11: Comparison: Tolvaptan; Statistical analysis at Week 94; Test type: Superiority or Other; p = 0.1346, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 12: Comparison: Tolvaptan; Statistical analysis at Week 106; Test type: Superiority or Other; p = 0.5237, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 13: Comparison: Tolvaptan; Statistical analysis at Week 118; Test type: Superiority or Other; p = 0.3476, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 14: Comparison: Tolvaptan; Statistical analysis at Week 130; Test type: Superiority or Other; p = 0.2488, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 15: Comparison: Tolvaptan; Statistical analysis at Week 142; Test type: Superiority or Other; p = 0.1598, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 16: Comparison: Tolvaptan; Statistical analysis at Week 154; Test type: Superiority or Other; p = 0.2820, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 17: Comparison: Tolvaptan; Statistical analysis at Week 166; Test type: Superiority or Other; p = 0.3743, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 18: Comparison: Tolvaptan; Statistical analysis at Week 178; Test type: Superiority or Other; p = 0.3600, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 19: Comparison: Tolvaptan; Statistical analysis at Week 190; Test type: Superiority or Other; p = 0.3101, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 20: Comparison: Tolvaptan; Statistical analysis at Week 202; Test type: Superiority or Other; p = 0.0269, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 21: Comparison: Tolvaptan; Statistical analysis at Week 214; Test type: Superiority or Other; p = 0.0944, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned

14. Secondary Outcome: Mean Change From Baseline in SF-12 (Health Survey) Physical Component Summary (PCS)
Description: The PCS assess the physical and mental dimensions of health-related quality of life. The PCS is equal to the sum of the items of endurance activities, strength activities, gross coordination activities, and fine coordination activities. The PCS is a computed score with weighted function based on the 12 questions from the 8 subscales (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, mental health) of the SF-12v1 questionnaire per instructions by the scale's publisher. The scale ranges from 0 to 100 with 0 representing the lowest level of health and 100 indicating the highest level of health.
Time Frame: Baseline to Week 214
Population: The ITT dataset comprised of data from all enrolled participants who had observations at Baseline and at least one Post-Baseline visit were analyzed. In the last observation carried forward (LOCF) dataset, missing data were filled in using the participant's preceding non-missing value, except that Baseline value will not be carried forward.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tolvaptan
Number analyzed (Participants) | 111
Units on a scale
  Day 14 (N= 102) | 1.0 (7.3)
  Day 31 (N= 106) | 0.4 (7.9)
  Week 10 (N= 106) | 0.3 (8.1)
  Week 18 (N= 106) | 0.4 (8.1)
  Week 26 (N= 106) | -0.9 (9.7)
  Week 34 (N= 106) | -0.3 (9.4)
  Week 42 (N= 106) | -1.1 (9.4)
  Week 50 (N= 106) | -1.1 (9.0)
  Week 58 (N= 106) | -0.9 (9.0)
  Week 70 (N= 106) | -1.1 (9.1)
  Week 82 (N= 106) | -0.9 (8.9)
  Week 94 (N= 106) | -1.6 (9.1)
  Week 106 (N= 106) | -1.7 (8.4)
  Week 142 (N= 2) | -9.1 (10.8)
  Week 166 (N= 2) | 4.6 (9.7)
  Week 178 (N= 2) | -11.3 (2.5)
  Week 190 (N= 6) | -2.2 (5.6)
  Week 202 (N= 1) | 0.6 (NA) — Standard deviation (SD) is not calculated at Week 202 as there was only 1 participant.
  Week 214 (N= 6) | 4.0 (9.2)
Statistical Analysis 1: Comparison: Tolvaptan; Statistical analysis at Day 14; Test type: Superiority or Other; p = 0.1739, Student t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 2: Comparison: Tolvaptan; Statistical analysis at Day 31; Test type: Superiority or Other; p = 0.6095, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 3: Comparison: Tolvaptan; Statistical analysis at Week 10; Test type: Superiority or Other; p = 0.6902, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 4: Comparison: Tolvaptan; Statistical analysis at Week 18; Test type: Superiority or Other; p = 0.6340, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 5: Comparison: Tolvaptan; Statistical analysis at Week 26; Test type: Superiority or Other; p = 0.3210, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 6: Comparison: Tolvaptan; Statistical analysis at Week 34; Test type: Superiority or Other; p = 0.7787, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 7: Comparison: Tolvaptan; Statistical analysis at Week 42; Test type: Superiority or Other; p = 0.2198, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 8: Comparison: Tolvaptan; Statistical analysis at Week 50; Test type: Superiority or Other; p = 0.1926, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 9: Comparison: Tolvaptan; Statistical analysis at Week 58; Test type: Superiority or Other; p = 0.3109, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 10: Comparison: Tolvaptan; Statistical analysis at Week 70; Test type: Superiority or Other; p = 0.2269, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 11: Comparison: Tolvaptan; Statistical analysis at Week 82; Test type: Superiority or Other; p = 0.2749, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 12: Comparison: Tolvaptan; Statistical analysis at Week 94; Test type: Superiority or Other; p = 0.0702, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 13: Comparison: Tolvaptan; Statistical analysis at Week 106; Test type: Superiority or Other; p = 0.0412, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 14: Comparison: Tolvaptan; Statistical analysis at Week 142; Test type: Superiority or Other; p = 0.4448, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 15: Comparison: Tolvaptan; Statistical analysis at Week 166; Test type: Superiority or Other; p = 0.6233, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 16: Comparison: Tolvaptan; Statistical analysis at Week 178; Test type: Superiority or Other; p = 0.1001, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 17: Comparison: Tolvaptan; Statistical analysis at Week 190; Test type: Superiority or Other; p = 0.3739, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 18: Comparison: Tolvaptan; Statistical analysis at Week 214; Test type: Superiority or Other; p = 0.3334, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned

15. Secondary Outcome: Mean Change From Baseline in SF-12 (Health Survey) Mental Component Summary (MCS)
Description: The MCS assess the physical and mental dimensions of health-related quality of life. The MCS is equal to the sum of the items of concentration activities, calculating activities, language activities, and memory activities. The MCS is a computed score with weighted function based on the 12 questions from the 8 subscales (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, mental health) of the SF-12v1 questionnaire per instructions by the scale's publisher. The scale ranges from 0 to 100 with 0 representing the lowest level of health and 100 indicating the highest level of health.
Time Frame: Baseline to Week 214
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tolvaptan
Number analyzed (Participants) | 103
Units on a scale
  Day 14 (N= 102) | -1.0 (8.8)
  Day 31 (N= 106) | -1.0 (9.6)
  Week 10 (N= 106) | -0.4 (9.8)
  Week 18 (N= 106) | -2.0 (8.8)
  Week 26 (N= 106) | -1.1 (8.8)
  Week 34 (N= 106) | -2.7 (9.4)
  Week 42 (N= 106) | -2.1 (10.1)
  Week 50 (N= 106) | -1.9 (10.4)
  Week 58 (N= 106) | -2.5 (11.4)
  Week 70 (N= 106) | -2.6 (10.7)
  Week 82 (N= 106) | -2.5 (10.5)
  Week 94 (N= 106) | -2.6 (10.5)
  Week 106 (N= 106) | -3.7 (11.6)
  Week 142 (N= 2) | -11.2 (27.6)
  Week 166 (N= 2) | 5.0 (13.6)
  Week 178 (N= 2) | 0.4 (4.5)
  Week 190 (N= 6) | -2.8 (8.2)
  Week 202 (N= 1) | -0.8 (NA) — SD was not calculated at Week 202 as there was only 1 participant.
  Week 214 (N= 6) | -0.5 (7.8)
Statistical Analysis 1: Comparison: Tolvaptan; Statistical analysis at Day 14; Test type: Superiority or Other; p = 0.2575, Student t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 2: Comparison: Tolvaptan; Statistical analysis at Day 31; Test type: Superiority or Other; p = 0.2715, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 3: Comparison: Tolvaptan; Statistical analysis at Week 10; Test type: Superiority or Other; p = 0.6860, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 4: Comparison: Tolvaptan; Statistical analysis at Week 18; Test type: Superiority or Other; p = 0.0224, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 5: Comparison: Tolvaptan; Statistical analysis at Week 26; Test type: Superiority or Other; p = 0.1871, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 6: Comparison: Tolvaptan; Statistical analysis at Week 34; Test type: Superiority or Other; p = 0.0039, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 7: Comparison: Tolvaptan; Statistical analysis at Week 42; Test type: Superiority or Other; p = 0.0325, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 8: Comparison: Tolvaptan; Statistical analysis at Week 50; Test type: Superiority or Other; p = 0.0631, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 9: Comparison: Tolvaptan; Statistical analysis at Week 58; Test type: Superiority or Other; p = 0.0277, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 10: Comparison: Tolvaptan; Statistical analysis at Week 70; Test type: Superiority or Other; p = 0.0128, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 11: Comparison: Tolvaptan; Statistical analysis at Week 82; Test type: Superiority or Other; p = 0.0164, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 12: Comparison: Tolvaptan; Statistical analysis at Week 94; Test type: Superiority or Other; p = 0.0119, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 13: Comparison: Tolvaptan; Statistical analysis at Week 106; Test type: Superiority or Other; p = 0.0013, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 14: Comparison: Tolvaptan; Statistical analysis at Week 142; Test type: Superiority or Other; p = 0.6691, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 15: Comparison: Tolvaptan; Statistical analysis at Week 166; Test type: Superiority or Other; p = 0.6923, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 16: Comparison: Tolvaptan; Statistical analysis at Week 178; Test type: Superiority or Other; p = 0.9292, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 17: Comparison: Tolvaptan; Statistical analysis at Week 190; Test type: Superiority or Other; p = 0.4401, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned
Statistical Analysis 18: Comparison: Tolvaptan; Statistical analysis at Week 214; Test type: Superiority or Other; p = 0.3609, Student's t-test — Descriptive use only, no statistical adjustments for multiplicity were planned

16. Secondary Outcome: Change From Baseline in the Hyponatremia Disease-specific Survey
Description: Analysis of individual items of Hyponatremia Disease-specific Survey was not conducted, because the analysis of Hyponatremia Disease-specific Survey was focused on the PCS and MCS summary scores since these 2 scores were developed. Subgroup analyses of Hyponatremia Disease-specific Survey were also not conducted.
Time Frame: Baseline to Week 214
Population: The Hyponatremia Disease-specific Survey PCS and MCS scores evaluated during the trial were variable with only nominal changes from baseline observed. The data were collected under 2 different datasets, so the number of participants in each dataset was reduced that limited analysis of this endpoint.
Arm/Group | Tolvaptan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs are reported from the signing of the informed consent until the follow-up visit (+7 days) after the last dose of study drug as scheduled or as an early termination.
Arm/Group | Tolvaptan
Serious Adverse Events (participants affected / at risk) | 76/111
Other Adverse Events (participants affected / at risk) | 86/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (N=111)
Anemia (Blood and lymphatic system disorders) | 4
Spontaneous haematoma (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 3
Atrial flutter (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 7
Cardiac failure congestive (Cardiac disorders) | 7
Cardiac tamponade (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 3
Left ventricular failure (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Goitre (Endocrine disorders) | 1
Blindness (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Retinal haemorrhage (Eye disorders) | 1
Retinoschisis (Eye disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 5
Colitis ischaemic (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Diverticulum (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastritis erosive (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5
Haematemesis (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Malaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Umbilical hernia perforation (Gastrointestinal disorders) | 1
Volvulus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Adverse drug reaction (General disorders) | 1
Chest pain (General disorders) | 5
Gait disturbance (General disorders) | 1
General physical health deterioration (General disorders) | 1
Hernia (General disorders) | 1
Multi-organ failure (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 1
Ulcer haemorrhage (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 2
Portal hypertensive gastropathy (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 2
Catheter site infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Clostridium difficile colitis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 1
Diabetic gangrene (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Heliobacter gastritis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Peritonitis bacterial (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 10
Sepsis (Infections and infestations) | 2
Sepsis syndrome (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 3
Urosepsis (Infections and infestations) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Hip fracture (Injury, poisoning and procedural complications) | 3
Humerus fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 2
Ulna fracture (Injury, poisoning and procedural complications) | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Troponin increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Failure to thrive (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypervolaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma unspecified histology aggressive refracto (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Altered state of consciousness (Nervous system disorders) | 1
Anoxic encephalopathy (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Dysphasia (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 5
Epilepsy (Nervous system disorders) | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 2
Hydrocephalus (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Reversible ischaemic neurological deficit (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Transient ischaemic attack (Nervous system disorders) | 2
Alcoholism (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Mental status changes (Psychiatric disorders) | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 1
Panic disorder (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Bladder neck sclerosis (Renal and urinary disorders) | 1
Hypertonic bladder (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 4
Renal failure acute (Renal and urinary disorders) | 3
Renal impairment (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Arteriosclerosis (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Lymphocele (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
Temporal arteritis (Vascular disorders) | 1
Vascular insufficiency (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (N=111)
Anaemia (Blood and lymphatic system disorders) | 16
Hypothyroidism (Endocrine disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 7
Ascites (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 20
Dyspepsia (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 10
Asthenia (General disorders) | 6
Chest pain (General disorders) | 8
Fatigue (General disorders) | 15
Oedema (General disorders) | 6
Oedema peripheral (General disorders) | 25
Pain (General disorders) | 6
Pyrexia (General disorders) | 6
Thirst (General disorders) | 14
Bronchitis (Infections and infestations) | 8
Gastroenteritis (Infections and infestations) | 7
Nasopharyngitis (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 18
Contusion (Injury, poisoning and procedural complications) | 8
Fall (Injury, poisoning and procedural complications) | 6
Skin laceration (Injury, poisoning and procedural complications) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 13
Hyponatraemia (Metabolism and nutrition disorders) | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10
Dizziness (Nervous system disorders) | 12
Headache (Nervous system disorders) | 15
Lethargy (Nervous system disorders) | 6
Insomnia (Psychiatric disorders) | 9
Pollakiuria (Renal and urinary disorders) | 12
Renal failure (Renal and urinary disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Ecchymosis (Skin and subcutaneous tissue disorders) | 7
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No